CLINICAL TRIAL: NCT05719636
Title: Effects of Progressive Resistance Exercise Training on Endurance and Functional Mobility in Children With Spina Bifida
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0740
Record Dates: First submitted 2023-01-31; First posted 2023-02-09 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Spina Bifida
Keywords: resistance exercise; endurance; functional mobility
MeSH Terms: conditions — Spinal Dysraphism

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator)
  Interventions: Other: Conventional treatment
- Progressive resistance exercise (Experimental)
  Interventions: Other: Progressive resistance exercise

INTERVENTIONS:
Other: Conventional treatment — Conventional protocol that involves simple active and passive range of motion exercises of lower limb with positioning for assistive devices was provided
  Arms: Conventional treatment
Other: Progressive resistance exercise — The protocol that was applied on the members of (experimental group) are progressive resistance exercises. These passive resistance exercises included Flexion, Extension, Abduction, Adduction of hip; Flexion, Extension of knee; with minimum time in start and minimum quantity of loads, with Thera bands and sandbags,.
  Arms: Progressive resistance exercise

SUMMARY:
In this research the effects of progressive resistance exercise training on endurance and functional mobility in children with spina bifida are assessed.

ELIGIBILITY:
Inclusion Criteria:

* 8 to 16 year.
* Male and female both are included.
* Lower extremity weakness (less than 2).
* Knee and hip flexion contractures

Exclusion Criteria:

* Bowel and bladder dysfunction.
* Children having absent tone.
* Children having bone fracture

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2022-05-13 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-04-20 (Actual)

PRIMARY OUTCOMES:
Patient Specific Functional Scale for lower extremity functional status | 6th week
  Patient Specific Functional Scale (PSFS) was developed by Stratford et al 1995 as a self-report outcome measure of function that could be used in patients with varying levels of independence. The aim of PSFS is to provide clinicians with a valid, reliable, responsive and efficient outcome measure that would be easy to use and applicable to a large number of clinical presentations. Gives the patient positive re-enforcement that the intervention is effective. Can be used on a wide variety of musculoskeletal and neurological conditions

SECONDARY OUTCOMES:
6 minute walk test | 6th week
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
sit to stand test | 6th Week
  The participant is encouraged to complete as many full stands as possible within 30 seconds. The participant is instructed to fully sit between each stand. While monitoring the participant's performance to ensure proper form, the tester silently counts the completion of each correct stand

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, MS, Principal Investigator — Riphah International University
Locations (1):
- Children hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No